CLINICAL TRIAL: NCT03398174
Title: Motor Control Exercise and Patient Education for the Management of Chronic Low Back Pain in a Low-Resource Rural Nigerian Community: A Pilot Randomized Controlled Trial.
Brief Title: A Pilot Study of Motor Control Exercise and Patient Education for the Management of Chronic Low Back Pain in Rural Nigerian Community.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Aminu A. Ibrahim, Doctoral Student, Bayero University Kano, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPS/PPT/15/00009
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Chronic Low Back Pain
Keywords: Rural dwellers; Patient Education; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participants' treatment allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Control Exercise Plus Patient Education (Experimental): Participants will receive a total of 12 sessions (2 sessions per week) of exercise program consisting of motor control training and group patient education session once a week (6 sessions) all over 6-weeks.
  The motor control training will be aiming at improving function of specific muscles of the lumbopelvic region and the control of posture and movement.
  The patient education program will be aiming to provide non-threatening information to enable patients to better understand their pain, change any unhelpful beliefs about LBP, and integrate self-management and active coping strategies that deals with fear avoidance behavior and catastrophic thought.
  In addition, participants will also perform stretching exercises and instructed to perform continuous overground walk.
  Interventions: Behavioral: Motor Control Exercise; Behavioral: Patient Education
- Motor Control Exercise (Experimental): Participants will receive the same motor control exercise program described in the patient education and motor control exercise group.
  In addition, participants will also perform stretching exercises and instructed to perform continuous overground walk.
  Interventions: Behavioral: Motor Control Exercise
- Patient Education (Experimental): Participants will receive the same patient education program described in the motor control exercise plus patient education group.
  In addition, participants will also perform stretching exercises and instructed to perform continuous overground walk.
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Motor Control Exercise — Exercise aiming at improving function of specific muscles of the lumbopelvic region and the control of posture and movement.
  In addition, participants will perform stretching exercises aiming at targeting the postural muscles and connective tissue around the lower back, pelvis and lower limb that tend to get shortened in chronic LBP, and they will be advised to perform aerobic exercise in the form of overground walking at desirable speed at home.
  Other Names: Specific Stabilisation Exercise
  Arms: Motor Control Exercise; Motor Control Exercise Plus Patient Education
Behavioral: Patient Education — Patient education to enable patients to better understand their pain, change any unhelpful beliefs about LBP, and integrate self-management and active coping strategies that deals with fear avoidance behavior and catastrophic thought.
  In addition, participants will perform stretching exercises aiming at targeting the postural muscles and connective tissue around the lower back, pelvis and lower limb that tend to get shortened in chronic LBP, and they will be advised to perform aerobic exercise in the form of overground walking at desirable speed at home.
  Other Names: Psychosocial Education
  Arms: Motor Control Exercise Plus Patient Education; Patient Education

SUMMARY:
The main purpose of this pilot single-blind randomized clinical trial is to assess the feasibility of implementing motor control exercise and patient education for the management of chronic low back pain (CLBP) in a low resource rural Nigerian community.

DETAILED DESCRIPTION:
This study will determine whether supervised exercise training emphasizing motor control exercise (MCE) approach and a designed patient education (PE) program based on the psychosocial approach will be feasible and acceptable in reducing pain intensity and functional disability among rural dwellers with CLBP in Nigeria.

Participants will be recruited and assigned to one of three intervention groups that include MCE group, PE group, or MCE plus PE gr using a simple random technique based on an electronic randomization table generated by a computer software program. Blinded assessment of all clinical outcomes will be performed at baseline and 6 weeks after randomization.

Primary outcomes include pain intensity and functional disability while secondary outcomes include overall treatment satisfaction.

Data will be analyzed using descriptive statistics, paired t-test, and ANOVA. All statistical analyses will be performed on SPSS (version 24.00) at an alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 65 years old.
* Primary complaint of LBP experienced at least over the previous 3-month duration.
* Ability to read/understand English or Hausa language.

Exclusion Criteria:

* Previous history of thoracic spine or lumbosacral spine surgery.
* Any neurological findings indicating radiculopathy.
* Evidence of serious spine pathology (e.g. tumor, infection, fracture, spinal stenosis, inflammatory disease).
* Unstable or severe disabling chronic cardiovascular and pulmonary disease.
* History of serious psychological or psychiatric illness.
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change in pain Intensity | Baseline and 6 weeks after beginning treatment.
  Pain Intensity will be measured by an 11-point (0-10) Numerical Pain Rating Scale (NPRS).
Change in functional disability | Baseline and 6 weeks after beginning treatment.
  Functional disability will be measured by Oswestry disability index (ODI). The questionnaire consists of 10 items with each item having six statements. All scores are summed, then multiplied by two to obtain the index (range 0 to 100) with higher score indicating greater disability.

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks after beginning treatment.
  Patient satisfaction with treatment will be assessed using a 5-point Likert scale ranging from "very dissatisfied" (0) to "very satisfied" (4), with higher scores reflecting greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Aminu A Ibrahim, BPT, MPT, Principal Investigator — Physiotherapy Department, Faculty of Allied Health Sciences, Bayero University, Kano. Nigeria
Locations (1):
- Tsakuwa Primary Healthcare Center, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim AA, Akindele MO, Ganiyu SO. Motor control exercise and patient education program for low resource rural community dwelling adults with chronic low back pain: a pilot randomized clinical trial. J Exerc Rehabil. 2018 Oct 31;14(5):851-863. doi: 10.12965/jer.1836348.174. eCollection 2018 Oct. PMID 30443533